CLINICAL TRIAL: NCT07265284
Title: A Phase Ⅰ/Ⅲ Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Picankibart in Adolescent Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate Efficacy and Safety of IBI112 in Adolescent Participants With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biopharmaceutical Technology (Hangzhou) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112A304
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Participants receive placebo through week 16,placebo participants will cross over to receive IBI112 through week 44
  Interventions: Drug: placebo
- IBI112 (Experimental): Participants receive IBI112 through week 44
  Interventions: Drug: IBI112

INTERVENTIONS:
Drug: IBI112 — IBI112 by subcutaneous injection
  Arms: IBI112
Drug: placebo — placebo by subcutaneous injection
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IBI112 in the treatment of adolescent participants with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Males or females aged 12 to 18 years; Diagnosed with plaque psoriasis and a history of psoriasis ≥6 months; suitable for phototherapy and/or systemic treatment for psoriasis.

Exclusion Criteria:

History of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease Participant has history of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis Has received any therapeutic agent directly targeted to IL-17within 6 months of the first administration of study agent Has received any therapeutic agent directly targeted toTNF-a within 3 months of the first administration of study agent Has received any conventional therapeutic agent within 1 months of the first administration of study agent Has received any topic therapeutic agent within 2 weeks of the first administration of study agent Hsa received IBI112

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and severity index(PASI) 75 at week 16 | week 16
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients achieving an static Physician's Global Assessment (sPGA) Score of Cleared (0) or Minimal (1) at Week 16 | week 16
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall.

SECONDARY OUTCOMES:
Percentage of patients achieving PASI 50 at week 16 | week 16
  PASI 50 is defined as at least a 50% reduction in PASI relative to baseline
Percentage of patients achieving PASI 90 at week 16 | week 16
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline
Percentage of patients achieving PASI 100 at week 16 | week 16
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients achieving an sPGA 0 at week 16 | week 16
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall.
Percentage of patients achieving an Children Dermatology life quality index (CDLQI) Score of 0 /1at week 16 | week 16
  The CDLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life
Percentage of patients achieving PASI 75 at week 56 | week 56
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients achieving PASI 90 at week 56 | week 56
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline
Percentage of patients achieving PASI 100 at week 56 | week 56
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients achieving an sPGA 0/1 at Week 56 | week 56
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall.
Percentage of patients achieving an sPGA 0 at Week 56 | week 56
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China